CLINICAL TRIAL: NCT04697667
Title: The Combination of Exercise and PRP vs Exercise Alone in Patients With Knee Osteoarthritis: A Randomized Controlled Clinical Trial
Brief Title: Exercise and PRP vs Exercise Alone in Patients With Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Sezen Karaborklu Argut, Researcher, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TDK-2020-35062
Record Dates: First submitted 2021-01-03; First posted 2021-01-06 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Double
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group I (Experimental): Each subject in this group will receive a combined treatment protocol consisting of three PRP injections to knee joint and supervised exercise program.
  Interventions: Other: Exercise; Biological: PRP
- Group II (Active Comparator): Each subject in this group will receive a treatment of supervised exercise program.
  Interventions: Other: Exercise
- Group III (Active Comparator): Each subject in this group will receive a treatment of three PRP injections to knee joint.
  Interventions: Biological: PRP

INTERVENTIONS:
Other: Exercise — Supervised exercise program
  Arms: Group I; Group II
Biological: PRP — Intra-articular PRP injections to knee joint
  Arms: Group I; Group III

SUMMARY:
This study is a prospective randomized controlled study of different treatments for knee osteoarthritis and aims to investigate the efficacy of exercise combined platelet rich plasma (PRP) injection versus only exercise or only PRP treatments.

ELIGIBILITY:
Inclusion Criteria:

* Adults 40-70 years of age,
* Grade 2-3 according to Kellgren Lawrence osteoarthritis classification,
* No medication for knee osteoarthritis in the past three months,
* Subjects who understand and sign the consent form for this study.

Exclusion Criteria:

* Patients who have received an invasive procedure, intra-articular application and / or physiotherapy in the target knee within three months,
* Previous partial or total knee replacement of the target knee,
* Body mass index > 30 kg/m2,
* Having any cardiovascular diseases, neurological disorders, rheumatic diseases, malignancy or psychiatric diseases,
* Impaired cognition that impacts the ability to give informed consent,
* Participation in another clinical trial.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2021-01-31 (Actual); Primary Completion 2022-01-07 (Actual); Study Completion 2022-02-10 (Actual)

PRIMARY OUTCOMES:
Pain intensity | 6th week
  Pain intensity will be measured using the numerical pain rating scale. Patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Pain intensity | 3rd month
  Pain intensity will be measured using the numerical pain rating scale. Patients are asked to circle the number between 0 and 10 that fits best to their pain intensity. Zero usually represents 'no pain at all' whereas the upper limit represents 'the worst pain ever possible'.
Function | 6th week
  Functional status of the patients will be evaluated by The Western Ontario and McMaster Universities Arthritis (WOMAC) Index. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales (Pain, Stiffness and Physical Function). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Higher scores on the WOMAC indicate worse results.
Functional performance - 40m fast-paced walk test | 6th week
  Functional performance of the patients will be evaluated by 40-meter fast-paced walk test. Participants are asked to walk as quickly but as safely as possible, without running, along a 10-meter walkway for a total distance of 40 meters. Walking speed will be measured in meters/second (m/s).
Functional performance - 10-step stair-climb test | 6th week
  Functional performance of the patients will be evaluated by 10-step stair-climb test. Patients are instructed to ascend and descend the flight of stairs as quickly as possible but in a safe manner. The time needed is recorded in seconds.
Function | 3rd month
  Functional status of the patients will be evaluated by The Western Ontario and McMaster Universities Arthritis (WOMAC) Index. It is a self-administered questionnaire consisting of 24 items divided into 3 subscales (Pain, Stiffness and Physical Function). The test questions are scored on a scale of 0-4, which correspond to: None (0), Mild (1), Moderate (2), Severe (3), and Extreme (4). Higher scores on the WOMAC indicate worse results.
Functional performance - 40m fast-paced walk test | 3rd month
  Functional performance of the patients will be evaluated by 40-meter fast-paced walk test. Participants are asked to walk as quickly but as safely as possible, without running, along a 10-meter walkway for a total distance of 40 meters. Walking speed will be measured in meters/second (m/s).
Functional performance - 10-step stair-climb test | 3rd month
  Functional performance of the patients will be evaluated by 10-step stair-climb test. Patients are instructed to ascend and descend the flight of stairs as quickly as possible but in a safe manner. The time needed is recorded in seconds.

SECONDARY OUTCOMES:
Range of motion | 6th week
  Knee joint ROMs will be measured using a universal goniometer. The process will be repeated three times and the average value will be recorded.
Range of motion | 3rd month
  Knee joint ROMs will be measured using a universal goniometer. The process will be repeated three times and the average value will be recorded.
Health related quality of life | 6th week
  Health related quality of life will be measured using SF 12 score that measures eight health domains to assess physical and mental health.
Health related quality of life | 3rd month
  Health related quality of life will be measured using SF 12 score that measures eight health domains to assess physical and mental health.
Patient Satisfaction | 6th week
  Patient satisfaction will be assessed by the Global Rating of Change scale.
Patient Satisfaction | 3rd month
  Patient satisfaction will be assessed by the Global Rating of Change scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)